CLINICAL TRIAL: NCT03784599
Title: Trastuzumab-emtansine and Osimertinib Combination Treatment to Target HER2 Bypass Track Resistance in EGFR Mutation Positive NSCLC
Brief Title: T-DM1 and Osimertinib Combination Treatment to Target HER2 Bypass Track Resistance in EGFR Mutation Positive NSCLC
Acronym: TRAEMOS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: insufficient effectiveness
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: AstraZeneca (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M18TEO
Record Dates: First submitted 2018-10-31; First posted 2018-12-24 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Ado-Trastuzumab Emtansine; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trastuzumab-emtansine and osimertinib (Experimental): Trastuzumab-emtansine 3.6 mg/kg, intravenously, every 3 weeks
  Osimertinib 80 mg once daily, orally, continuous
  Treatment will be continued until tumor progression (according to RECIST v1.1) confirmed by tumor imaging, unacceptable toxicity, or death occurs.
  Interventions: Drug: Trastuzumab emtansine; Drug: Osimertinib

INTERVENTIONS:
Drug: Trastuzumab emtansine — Infusion
Drug: Osimertinib — Tablet

SUMMARY:
This is a single arm open-label multi-center phase II study, investigating disease control rate after 3 months of treatment with trastuzumab-emtansine/osimertinib combination therapy in patients with advanced EGFR mutation positive non-small cell lung cancer (NSCLC) with HER2 bypass track resistance.

DETAILED DESCRIPTION:
This study is a multicenter single arm phase II study with a phase I run in to study the toxicity and efficacy of T-DM1 and osimertinib combination treatment in patients with EGFR mutated NSCLC and HER2 bypass track activation (HER2 immunohistochemistry (IHC) ≥2+ and/or HER2 amplification) after progression on an EGFR TKI.

In the phase I run in, study safety will be assessed in a classical 3+3 design. Because of potential for overlapping hematologic and non-hematologic adverse events (AE), the first 3 patients will receive a reduced dose of T-DM1 3.0 mg/kg IV every 3 weeks combined with osimertinib 80 mg once daily. Dose-limiting toxicity (DLT) is defined as a grade 3 AE toxicity according to CTC AE 4.03 that does not recover to grade ≤2 before the next cycle of T-DM1. DLT's will be collected up to 6 weeks after treatment initiation (2 T-DM1 cycles). Dose escalation within patients is not allowed.

If 1 patient develops a dose-limiting toxicity (DLT), 3 more will be included and treated with T-DM1 3.0 mg/kg. If ≥2 of the 6 patients develop a DLT, further study of the combination will be halted. Otherwise, T-DM1 3.0 mg/kg IV every 3 weeks combined with osimertinib 80 mg once daily will be the maximum tolerated dose (MTD) to put forward in the phase II part of this study.

If none of the first three patients develops a DLT, the T-DM1 dose will be escalated to the standard dose of 3.6 mg/kg. If ≤1 patient experiences a DLT in 6 patients (3+3), T-DM1 3.6 mg/kg IV every 3 weeks and osimertinib 80 mg once daily will be the MTD. If ≥2 patients develop a DLT, the T-DM1 will be lowered to 3.0 mg/kg and three more patients will be enrolled in this dose cohort. When ≤1 of these patients develops a DLT, this will be the MTD.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed stage IV non-squamous NSCLC, characterized by an activating EGFR mutation.
2. Progressive disease according to RECIST 1.1 on first (gefitinib, erlotinib), second (afatinib) or third (osimertinib) generation EGFR TKI and still receiving the drug.
3. A rebiopsy after having acquired resistance to a first, second or third generation TKI-treatment must have been performed and be:

   1. Negative for T790M in case of treatment with a first or second generation EGFR TKI. After progression on a third generation EGFR TKI patients may either be positive or negative for T790M.
   2. Positive for HER2-overexpression (positive membranous immunohistochemistry staining IHC ≥2+ (on a scale of 0-3) in ≥10% of the cells) must have been detected.
4. There must be at least one measurable disease site, according to RECIST 1.1 criteria.

   Patients need At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements.
5. Absence of symptomatic brain metastases. All patients will be scanned at baseline with a brain MRI.
6. Patients must be willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
7. World Health Organization (WHO) performance status 0-2.
8. Patients must have a life expectancy ≥12 weeks.
9. Ability to give written informed consent before patient screening.
10. Patients must be ≥18 years of age.
11. Men and women of child bearing potential should be willing to take adequate contraceptive measures during the study and until three months after study drug discontinuation

Exclusion Criteria:

1. Uncontrolled infectious disease.
2. Other active malignancy. Patients with a history of cancer for which treatment is complete and with no evidence of malignant disease currently cannot be enrolled if their chemotherapy was completed less than 6 months prior and/or have received a bone marrow transplant less than 2 years before the first day of study treatment.
3. Major surgery (excluding diagnostic procedures like e.g. mediastinoscopy or VATS biopsy) in the previous 4 weeks.
4. Known hypersensitivity to T-DM1 or osimertinib (or drugs with a similar chemical structure or class) or any excipients of these agents.
5. Previous treatment with a HER2 monoclonal antibody.
6. Clinically significant cardiac disease or:

   * Patients with pre-treatment LVEF < 55%.
   * Prior history of congestive cardiac failure; LVEF decline to <50% on previous treatment with HER2 agents
   * Conditions impairing LV function e.g. uncontrolled hypertension
   * MI/unstable angina within 6 months or serious cardiac arrhythmia
7. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (QTc) > 470 msec obtained from 3 electrocardiograms (ECGs), using the screening clinic ECG machine derived QTc value
   * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g. complete left bundle branch block, third degree heart block and second degree heart block.
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval.
8. Inadequate bone marrow reserve or organ function, as demonstrated by any of the following laboratory values:

   * Hematology: hemoglobin <5.6 mmol/L, absolute neutrophil count <1.5 x 10^9/L, platelet count <100 x 10^9/L.
   * Biochemistry: alanine aminotransferase, aspartate aminotransferase and bilirubin ≤ 2.5 x ULN, except in the case of liver metastases where these values must be ≤ 5x ULN.
   * Kidney function: serum creatinine >1.5 x ULN concurrent with creatinine clearance <50 ml/min (measured or calculated by Cockroft and Gault equation).
9. Patients with symptomatic central nervous system metastases who are neurologically unstable. Unstable brain metastases except for those who have completed definitive therapy and have had a stable neurological status for 2 weeks after completion of definitive therapy. Patients may be on corticosteroids to control brain metastases if they have been on a stable dose for 2 weeks prior to the start of study treatment and are clinically asymptomatic.
10. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow osimertinib or previous significant bowel resection that would preclude adequate resorption of osimertinib.
11. Males and females of reproductive potential who are not using an effective method of birth control and females who are pregnant or breastfeeding or have a positive (serum) pregnancy test prior to study entry.
12. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
13. Treatment with an investigational drug within five half-lives of the compound or 3 months, whichever is greater
14. Currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be potent inducers of CYP3A4 (at least 3 week prior) (Appendix C). All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on CYP3A4.
15. Any unresolved toxicities from prior therapy greater than CTCAE grade 1 at the time of starting study treatment, with the exception of alopecia and grade 2, prior platinum-therapy-related neuropathy.
16. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
17. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment or any evidence of clinically active interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
Safety (intensity and incidence of adverse events) | Up to 30 days after last study drug intake
  Safety as indicated by intensity and incidence of adverse events, graded according to NCI CTCAE Version 4.03
Objective response rate according to RECIST v1.1 after 3 months of treatment | From date of registration until 3 months.
  Complete response and partial response after 3 months of treatment

SECONDARY OUTCOMES:
Progression-free survival | From date of registration until the date of first documented progression up to 100 months
  PFS, defined as the time from first administration of the study drug combination to disease progression by RECIST v1.1. or lost to follow up or death, whichever comes first
Disease control rate, after 3 months of treatment | From date of registration until 3 months.
  DCR, defined as the percentage of patients with stable disease (SD), partial response (PR) or complete response (CR)
Overall survival | From date of registration until the date of death from any cause, assessed up to 100 months.
  OS, defined as the time from first administration of the study drug combination to lost to follow up or death, whichever comes first

OTHER OUTCOMES:
Genetic profiling to assess predictors of response and resistance - circulating free (cf)DNA | At baseline, every 6 weeks and at treatment discontinuation (expected 6 months after start)
  cfDNA samples will be collected to assess predictors of response and resistance

CONTACTS AND LOCATIONS:
Overall Officials: J. de Langen, MD, PhD, Principal Investigator — NKI-AvL
Locations (5):
- Netherlands (5):
  - Maastricht UMC+, Maastricht, Limburg
  - VU medical center, Amsterdam, North Holland
  - Antoni van Leeuwenhoek ziekenhuis - Netherlands Cancer Institute, Amsterdam, North Holland
  - Erasmus MC, Rotterdam, South Holland
  - Univercity Medical Center Groningen, Groningen

IPD SHARING:
Plan to Share IPD: Undecided